CLINICAL TRIAL: NCT02407678
Title: An Open Label Phase 2 Clinical Trial of Retinal Gene Therapy for Choroideremia Using an Adeno-associated Viral Vector (AAV2) Encoding Rab-escort Protein 1 (REP1)
Brief Title: REP1 Gene Replacement Therapy for Choroideremia
Acronym: REGENERATE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Moorfields Eye Hospital NHS Foundation Trust (Other); University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REGEN2015
Record Dates: First submitted 2015-03-10; First posted 2015-04-03 (Estimated); Last update posted 2021-08-05 (Actual); Status verified 2021-07

CONDITIONS: Choroideremia
MeSH Terms: conditions — Choroideremia

STUDY DESIGN:
Intervention Model Description: The decision about which eye to treat will be made on clinical grounds and will generally be the worse eye affected in cases where BCVA differs between the two eyes by 2 lines or more of ETDRS letters. The eye to be treated will be randomised in cases where the degeneration is relatively symmetrical between the two eyes, defined as:
  * a difference in BCVA of no more than 1 line of ETDRS letters, and
  * no more than 25% difference in the area of surviving RPE as measured by fundus autofluorescence.
  Prospective participants having non-symmetrical retinal degeneration will be allocated to the non-randomised arm. The treated eye will generally be the worse eye. Prospective participants having relatively symmetrical retinal degeneration will be allocated to the randomised arm.
Masking Description: The study is designated as Open Label with no masking. However, in order to minimise bias evaluation of the treated eye and untreated fellow eye (control eye), the ophthalmic assessments (visual acuity, microperimetry, fundus autofluorescence, etc.) will be conducted by an appropriately qualified masked observer once the participant's treated eye has had time to heal after the surgical procedure and has regained its normal appearance and function.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment (Experimental): Treated eye undergoes AAV-mediated REP1 gene replacement. AAV vector is delivered by subretinal injection.
  Interventions: Genetic: AAV-mediated REP1 gene replacement
- Control (No Intervention): Untreated eye

INTERVENTIONS:
Genetic: AAV-mediated REP1 gene replacement — AAV vector carrying human REP1 gene is delivered into the treated eye by subretinal injection
  Arms: Treatment

SUMMARY:
The assessment of the efficacy (with respect to preservation of visual function and retinal structure) and safety of a single subretinal injection of AAV2.REP1 in participants with a confirmed diagnosis of choroideremia, as evaluated by various functional and anatomical outcomes measured over a number of time points up to 24 months post-treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Candidate is willing and able to give informed consent for participation in the study.
2. Male aged 18 years or above.
3. Genetic or molecular confirmed diagnosis of choroideremia (REP1 protein deficiency).
4. Active disease visible clinically within the macula region.
5. Best corrected visual acuity better than or equal to 6/60 (20/200; Decimal 0.1; LogMAR 1.0) in the study eye.

Exclusion Criteria:

1. Any female, or a male aged below 18 years.
2. An additional cause for sight loss (e.g. amblyopia) in the eye to be treated.
3. Any other significant ocular and non-ocular disease or disorder which, in the opinion of the investigator, may put the participants at risk because of participation in the study.
4. Inability to take systemic prednisolone for a period of 45 days.
5. Unwillingness to use barrier contraception methods for a period of three months following gene therapy surgery.
6. Participation in another research study involving an investigational product in the preceding 12 weeks.

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-08-16 (Actual); Primary Completion 2021-07-23 (Actual); Study Completion 2021-07-23 (Actual)

PRIMARY OUTCOMES:
Change from baseline in best corrected visual acuity in the treated eye | 2 years

SECONDARY OUTCOMES:
Change from baseline in the central visual field in the treated eye as determined by microperimetry | 2 years
Change from baseline in the area of surviving retinal pigment epithelium in the treated eye as measured by fundus autofluorescence, compared to the untreated fellow eye (control eye) after randomisation of treatment to one eye or the other | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Robert E MacLaren, MB ChB DPhil, Principal Investigator — University of Oxford
Locations (2):
- United Kingdom (2):
  - Moorfields Eye Hospital NHS Foundation Trust, London
  - Oxford University Hospitals NHS Foundation Trust, Oxford